CLINICAL TRIAL: NCT04295278
Title: An Observational Phase 0 Study to Assess the Performance and Real-world Feasibility of Implementing the MicroKine Dx Biomarker-based Risk Stratification of Critically-ill Pediatric Patients
Brief Title: Feasibility Study of MicroKine Dx System in Critically-ill Pediatric Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PreDxion Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PDXN-BP-001
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Systemic inflammatory response syndrome: Systemic inflammatory response syndrome in patients in the pediatric intensive care unit.
  Interventions: Diagnostic Test: MicroKine Dx system

INTERVENTIONS:
Diagnostic Test: MicroKine Dx system — Biomarker concentrations will be determined using the MicroKine Dx system and results will be compared to measurements taken using standard immunoassays.

SUMMARY:
This study will enroll approximately 25 pediatric patients to assess the performance and real-world feasibility of multi-biomarker based prognostic and predictive algorithms to aid in the clinical management of pediatric critically-ill patients.

DETAILED DESCRIPTION:
This study will enroll approximately 25 pediatric patients to assess the predictive performance of multi-biomarker based prognostic and predictive algorithms to aid in the clinical management of pediatric critically-ill patients.

All enrolled patients will undergo a series of blood collection procedures during their admission to the pediatric intensive care unit. The levels of inflammatory cytokines, chemokines, and effectors will be assessed and used in multi-biomarker based prognostic and predictive algorithms to determine patients at risk of in-hospital mortality.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 38 weeks gestation to 21 years of age
2. Admitted to the PICU within the prior 24 hours
3. Indwelling catheters for obtaining blood
4. Meet ≥2 age-adapted SIRS criteria

Key Exclusion Criteria:

1. Anticipated pediatric intensive care unit admission <24 hours
2. Primary immunodeficiency
3. Limited resuscitation, no escalation of treatment, do not resuscitate, or other limitations to care

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 38 Weeks to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric critically-ill patients 38-weeks gestation to 21 years of age admitted to a pediatric intensive care unit within the last 24-hours, with >1 indwelling central catheter, and meeting ≥2 age-adapted SIRS criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28-day
  28-day in hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Information, Study Director — PreDxion Bio, Inc.

IPD SHARING:
Plan to Share IPD: Undecided